CLINICAL TRIAL: NCT04231305
Title: Complications in Skin Grafts When Continuing Antithrombotic Therapy Prior to Cutaneous Surgery Requiring Skin Grafting: an Observational Study
Brief Title: Antithrombotics and Complications in Skin Grafts
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Lene Birk-Sørensen, Post Doc in Clinical Nursing, Aalborg University Hospital
Other Study IDs: 2019-29-12
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Skin Graft Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients who were referred to cutaneous surgery and needed full thickness or split skin grafting and using antitrombotic or non-antitrombotic therapies were observed. Data on patient characteristics, diagnosis, location of surgery and surgery performed, antithrombotic medication and complications in skin grafts were collected. Skin grafts were traced on a transparent film and areas of unhealed skin graft were marked

DETAILED DESCRIPTION:
Use of anticoagulants is common and practice regarding continuation or discontinuation of the medication peri-operatively for cutaneous surgery lacks evidence-based consensus. Therefore, patients who were referred to cutaneous surgery and needed full thickness or split skin grafting and using antitrombotic or non-antitrombotic therapies were observed. Data on patient characteristics, diagnosis, location of surgery and surgery performed, antithrombotic medication and complications in skin grafts were collected. Skin grafts were traced on a transparent film and areas of unhealed skin graft were marked

ELIGIBILITY:
Inclusion Criteria:

Patients referred to cutanous surgery with full thickness or split skin grafting. The excision should be performed on the levels of subcutis or perichondrium -

Exclusion Criteria:

Patients having a pacemaker, needed skin graft on bare bone and patients with an INR above 3.5

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 172 patients (92 males and 80 females) having 187 skin grafts were included. Avarage size of the skin grafts were 1278 mm2 ranging from 52mm2 to 14283mm2. Skin grafts where the patients received no or paused antithrombotic treatment were 90 while 97 skin grafts belonged to patients in antithrombotic treatment
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding | 5-7 postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Lene Birk-Sørensen, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided